CLINICAL TRIAL: NCT03790540
Title: Pain Assessment During Mandibular Nerve Block Injection With the Aid of Dental Vibe Tool in Pediatric Dental Patients: A Randomized Controlled Trial.
Brief Title: Pain Assessment During Mandibular Nerve Block Injection With the Aid of Dental Vibe Tool in Pediatric Dental Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: DentalVibe during LA
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia, Local
Keywords: DentalVibe; Mandibular nerve block injection; Consolability Scale

STUDY DESIGN:
Intervention Model Description: Each group will receive 2 mandibular nerve block injections with two different injection techniques, with 1-2 weeks apart as a washing out period .Mandibular nerve block injection will be either with vibration using DentalVibe at the injection side or topical analgesic (benzocaine 20%) gel will be applied before the injection of local anesthesia at first the appointment, and the alternative technique will be used at the second appointment. Injection with the aid of DentalVibe tool will act as the experimental group while the control group will be the use of topical analgesic (benzocaine 20%).
Masking Description: The operator will not be blinded to the type of treatment. However, the statistician will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Injection with the aid of DentalVibe (Experimental): 1 mL of Mepivacaine HCl 2%, 1/20000 Levonordefrin will be injected using a 27 gauge dental needle.
  DentalVibe is a small, handheld cordless device that has a charging docking station. A demonstration of DentalVibe (DV) will be performed by putting it into direct contact with the children's nails before applying the device intraorally. Then, the device will be placed on the oral mucosa to enclose the injection site before administering local anesthesia and Potential subject-expectancy effects and pressure from the placement of DV will be controlled. The device will be turned on to stimulate the area of needle penetration. After 5 seconds of vibration, the needle will be inserted. The device will continue vibrating during needle insertion and anesthetic injection.
  Interventions: Device: DentalVibe
- Injection with topical benzocaine 20% (Active Comparator): Topical anesthesia -Benzocaine gel 20%. Tissues will be dried using (2 X 2) gauze to enhance the absorption of the benzocaine gel 20% around the site of the needle penetration and will be left in contact with the soft tissue for one minute. Then the local anesthetic solution (1 ml Mepivacaine HCl 2%, 1/20000 Levonordefrin) will be injected using a 27 gauge dental needle.
  Interventions: Drug: Topical Benzocaine 20%

INTERVENTIONS:
Device: DentalVibe — It is a vibrotactile device that aids in reducing pain during local anesthesia injection in pediatric patients
  Arms: Injection with the aid of DentalVibe
Drug: Topical Benzocaine 20% — Topical benzocaine 20% gel on the mucosal injection site prior to injection
  Arms: Injection with topical benzocaine 20%

SUMMARY:
The purpose of this study is to valuate the effectiveness of DentalVibe(DV) tool in pain reduction during local anesthetic injection compared to traditional injection without aid of DentalVibe in pediatric patients.

DETAILED DESCRIPTION:
This study is a crossover randomized controlled clinical trial where (N=60 ) children will be selected from the outpatient clinic of Pediatric Dentistry and Public Health Department, Faculty of Dentistry, Alexandria University after securing necessary consents. These children will be selected based on a need for local anesthesia for pulpotomy treatment on both sides of the mandible. All selected children will be randomly allocated into 2 groups. Group I (assigned to injection with the aid of DentalVibe tool), Group II(assigned to conventional injection). Each group will receive 2 mandibular nerve block injections with two different injection techniques, with 1-2 weeks apart as a washing out period. Mandibular nerve block injection will be either with vibration using DentalVibe at the injection side or topical analgesic (benzocaine 20%) gel will be applied before the injection of local anesthesia at first the appointment, and the alternative technique will be used at the second appointment . Injection with the aid of DentalVibe tool will act as the experimental group while the control group will be the use of topical analgesic (benzocaine 20%).

ELIGIBILITY:
Inclusion Criteria:

* Age range from 5-7 years.
* Patients who are in need of pulpotomy dental treatment requiring bilateral local anesthesia in the mandible.
* Children free of any systemic disease or special health care needs.
* Positive or definitely positive behavior during preoperative assessments according to the Frankl Scale.

Exclusion Criteria:

* Having active sites of pathosis in the area of injection that could affect anesthetic assessment.
* Signs of irreversible pulpitis or pulp necrosis.
* Radiographs show periapical or bifurcation radiolucency.
* Patients allergic to local anesthesia or having a family history of allergy to local anesthesia.
* Patients with acute oral or facial infection (swelling and/or cellulitis).
* Patients refusing to participate.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Subjective pain reduction during local anesthesia administration. | during administration of local anesthesia
  Pain will be assessed during local anesthesia injection by means of Wong-Baker faces scale. It consists of faces with different facial expression for happiness and pain and is scored from 0-5 as 0 is very happy and feels no pain and 5 is very painful
Objective pain assessment after local anesthesia administration | after performing all injections
  After performing all the injections, pain reaction will be evaluated by two investigators independently using recorded video tapes by Face, Leg, Activity, Cry, Consolability Scale (FLACC).
  The scale comprises the following parameters:
  (1) Face, (2) Legs, (3) Activity, (4) Cry, and (5) Consolability. Each of the five categories is scored from 0 to 2, which results in a minimum score of 0 and maximum of 10. According to this scale 0 = relaxed and comfortable (no pain), 1-3 = mild discomfort, 4-6 = moderate pain, and 7-10 = severe discomfort or pain, A lower score represents less physical reaction than does a higher number.

CONTACTS AND LOCATIONS:
Overall Officials: Passant H Hassanein, BDS, Principal Investigator — Alexandria University; Amani M Khalil, PhD, Study Director — Alexandria University; Dalia AM Talaat, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Sermet Elbay U, Elbay M, Yildirim S, Kaya E, Kaya C, Ugurluel C, BaydemIr C. Evaluation of the injection pain with the use of DentalVibe injection system during supraperiosteal anaesthesia in children: a randomised clinical trial. Int J Paediatr Dent. 2016 Sep;26(5):336-45. doi: 10.1111/ipd.12204. Epub 2015 Sep 15. PMID 26369274
- [Background] Hutchins HS Jr, Young FA, Lackland DT, Fishburne CP. The effectiveness of topical anesthesia and vibration in alleviating the pain of oral injections. Anesth Prog. 1997 Summer;44(3):87-9. PMID 9481967
- [Background] Ram D, Peretz B. The assessment of pain sensation during local anesthesia using a computerized local anesthesia (Wand) and a conventional syringe. J Dent Child (Chic). 2003 May-Aug;70(2):130-3. PMID 14528773
- [Background] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149